CLINICAL TRIAL: NCT05263284
Title: A Phase 1 Trial of 8-Chloro-Adenosine in Combination With Venetoclax in Patients With Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: 8-Chloroadenosine in Combination With Venetoclax for the Treatment of Patients With Relapsed/Refractory Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21380; NCI-2022-00234 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21380 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2022-02-08; First posted 2022-03-02 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia; Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — 8-chloroadenosine; beta-apocarotenoid-14',13'-dioxygenase; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (8-chloroadenosine, venetoclax) (Experimental): Patients receive 8-Cl-Ado IV over 4 hours daily on days 1-5 and venetoclax PO QD on days 1-28. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: 8-Chloroadenosine; Drug: Venetoclax

INTERVENTIONS:
Drug: 8-Chloroadenosine — Given IV
  Other Names: 8-Chloro-adenosine; 8-Cl-adenosine; 8-Cl-Ado
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of a new 8-chloroadenosine in combination with venetoclax in treating patients with acute myeloid leukemia that has come back (relapsed) or does not respond to treatment (refractory). 8-Chloroadenosine may help block the formation of growths that may become cancer. Venetoclax is in a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. It may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Giving 8-chloroadenosine in combination with venetoclax may help prevent the disease from coming back in patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the safety and tolerability of a regimen combining 8-chloro-adenosine (8-Cl-Ado) and venetoclax in patients with relapsed or refractory (R/R) acute myeloid leukemia (AML), including type, frequency, severity, attribution, and duration of the toxicity.

II. Establish the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of 8-Cl-Ado when given in combination with venetoclax.

SECONDARY OBJECTIVES:

I. Obtain preliminary estimates of the anti-leukemia activity of the 8-Cl-Ado/venetoclax regimen by assessing the overall response rate (Complete remission[CR]+ complete remission with incomplete hematologic recovery [CRi]+ partial response [PR]) and complete remission rate (CR+CRi).

II. Obtain preliminary estimates of duration of remission (DOR), overall survival (OS), and event-free survival (EFS).

III. Determine the pharmacokinetics (PK) of plasma 8-Cl-Ado and metabolites when 8-Cl-Ado is given in combination with venetoclax.

EXPLORATORY OBJECTIVES:

I. Evaluate PK and pharmacodynamics (PD) of VEN/8-Cl-Ado combination therapy to identify biomarkers of clinical response and resistance.

II. Identify genes and pathways associated with response to VEN/8-Cl-Ado. III. Determine the metabolic consequences of VEN/8 Cl-Ado treatment on leukemia stem cells (LSCs).

OUTLINE:

Patients receive 8-Cl-Ado intravenously (IV) over 4 hours daily on days 1-5 and venetoclax orally (PO) once daily (QD) on days 1-28. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 28 days for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative.
* Age: >= 18 years.
* Eastern Cooperative Oncology Group (ECOG) =< 2.
* Life expectancy > 3 months.
* Patients with histologically confirmed acute myeloid leukemia (AML), according to World Health Organization (WHO) criteria, with relapsed/refractory disease.
* Patients must have any one of the following treatment history criteria:

  * Relapsed AML

    * Failed at least 1 line of salvage therapy or
    * Untreated relapse and are not candidates for allogeneic hematopoietic stem cell transplantation (alloHCT)
  * De novo AML

    * have not achieved complete response (CR) after 2 lines of therapy or
    * refractory to frontline therapy and not eligible for alloHCT
  * AML evolving from myelodysplastic syndrome (MDS) or myeloproliferative disorder who have failed hypomethylating agents (HMA) or induction chemotherapy
  * Patients who have relapsed after allo-HCT are eligible if they are at least 3 months after HCT, do not have active graft versus host disease (GVHD) and are off immunosuppression except for maintenance dose of steroids (prednisone 10 mg/day or less).
* Male subjects must agree to not donate sperm while taking protocol therapy through at least 90 days after the last dose.
* White blood cell (WBC) =< 25 x 10^9/L prior to initiation of venetoclax. Cytoreduction with hydroxyurea prior to treatment and/or during cycle 1 may be required.
* Total bilirubin =< 1.5 X upper limit of normal (ULN) (unless has Gilbert's disease).
* Aspartate aminotransferase (AST) =< 2.5 x ULN.
* Alanine aminotransferase (ALT) =< 2.5 x ULN.
* Creatinine clearance of >= 50 mL/min per 24 hour urine test or the Cockcroft-Gault formula.
* QTc =< 480 ms.
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Agreement by females and males of childbearing potential* to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 6 months (females) and 3 months (males) after the last dose of protocol therapy.

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only).

Exclusion Criteria:

* Current or planned use of other investigational agents, antineoplastic, biological, chemotherapy, or radiation therapy during the study treatment period, or within 2 weeks prior to day 1 of protocol therapy, with the following exception:

  * Hydroxyurea which may be continued through cycle 1.
* Expected to undergo HCT within 120 days of enrollment.
* Current or planned use of agents that prolong or suspected to prolong QTc.
* Received strong or moderate CYP3A inducers or St. John's Wort within 7 days prior to day 1 of protocol therapy.
* Received strong or moderate CYP3A inhibitors, or consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or Star fruit within 3 days prior to day 1 of protocol therapy.
* P-glycoprotein (P-gp) inhibitors within 7 days prior to day 1 of protocol therapy.
* Narrow therapeutic index P-gp substrates within 7 days prior to day 1 of protocol therapy.
* Acute promyelocytic leukemia.
* Active central nervous system (CNS) leukemia.
* Active fungal infection or bacterial sepsis.
* Class III/IV cardiovascular disability according to the New York Heart Association classification.
* Participants with clinically significant arrhythmia or arrhythmias not stable on medical management within two weeks of enrollment. Subjects with controlled, asymptomatic atrial fibrillation can enroll.
* History of acute cardiovascular ischemic event, i.e., myocardial infarction or unstable angina within 6 months of enrollment.
* History of unexplained syncope, significant histories of CAD (requiring revascularization by percutaneous coronary intervention [PCI] or coronary artery bypass grafting [CABG]), cardiomyopathy (ejection fraction [EF] < 50%).
* Prior surgery or gastrointestinal dysfunction that may affect drug absorption (e.g., gastric bypass surgery, gastrectomy).
* Unable to swallow capsules, has a partial or small bowel obstruction, or has a gastrointestinal condition resulting in a malabsorptive syndrome (e.g. small bowel resection with malabsorption).
* Active peptic ulcer disease.
* Other active malignancy except for localized skin cancer, bladder, prostate, breast or cervical carcinoma in situ.
* Females only: Pregnant or breastfeeding.
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures.
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2029-01-25 (Estimated); Study Completion 2029-01-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 1 year
  Toxicities will be graded using the National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events version 5.0.
Dose limiting toxicity (DLT) | Up to 1 cycle (Each cycle is 28 days)
  Toxicities will be graded using the NCI-Common Terminology Criteria for Adverse Events version 5.0. DLT will be assessed after cycle one.

SECONDARY OUTCOMES:
Time to response | Up to 1 year
  Defined by European LeukemiaNet (ELN) criteria 2017 in response-evaluable participants that achieve a best response of either complete remission (CR), complete remission with incomplete hematologic recovery (CRi), or partial response (PR) at the end of study therapy. Will be estimated using the product-limit method of Kaplan and Meier.
Duration of response (DOR) | From the first achievement of PR, CR, or CRi to time of disease progression, assessed up to 1 year
  Patients will be considered evaluable for response if they are eligible, have baseline disease assessments, and receive 2 cycles of protocol treatment, or achieve a CR/CRi after 1 cycle of protocol treatment, or progressed. Patients will have their response classified according to the European Leukemia Network (ELN) 2017 criteria. Will be estimated using the product-limit method of Kaplan and Meier.
Overall survival (OS) | From start of protocol treatment to time of death due to any cause, or until last follow-up, assessed up to 1 year
  Patients will be considered evaluable for response if they are eligible, have baseline disease assessments, and receive 2 cycles of protocol treatment, or achieve a CR/CRi after 1 cycle of protocol treatment, or progressed. Patients will have their response classified according to the European Leukemia Network (ELN) 2017 criteria. Will be estimated using the product-limit method of Kaplan and Meier.
Event-free survival (EFS) | From start of protocol treatment to time of disease relapse/progression or death due to any cause, whichever occurs earlier; or until last follow-up, assessed up to 1 year
  Patients will be considered evaluable for response if they are eligible, have baseline disease assessments, and receive 2 cycles of protocol treatment, or achieve a CR/CRi after 1 cycle of protocol treatment, or progressed. Patients will have their response classified according to the European Leukemia Network (ELN) 2017 criteria. Will be estimated using the product-limit method of Kaplan and Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Vinod Pullarkat, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States